CLINICAL TRIAL: NCT00704717
Title: Evaluation of Satisfaction in Patients Receiving PegIntron Pen / Rebetol for Hepatitis C
Brief Title: Evaluation of Patient Satisfaction in Hepatitis C Patients Treated With PegIntron Pen and Rebetol in Romania (Study P04301)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04301
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; penclomedine; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Treated Patients: All patients participating in the study.
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031) pen; Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) pen — PegIntron pen administered in accordance with approved labeling
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered in accordance with approved labeling.
  Other Names: SCH 18908

SUMMARY:
The objective of this study is to evaluate patient satisfaction in hepatitis C patients receiving PegIntron pen plus Rebetol. The rationale is that the effectiveness of treatment is correlated with adherence to the prescribed regimen which, in turn, is affected by the ease of use and accuracy of treatment administration. Since the PegIntron pen is a novel device, the results of this study will be used to improve the training of patients and healthcare providers in PegIntron pen use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatitis C under treatment with PegIntron Pen and Rebetol in Romania.

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hepatitis C under treatment with PegIntron Pen plus Rebetol therapy at approximately 70 sites in Romania.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Treated Patients
Started | 185
Completed | 185
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Treated Patients
Number analyzed (Participants) | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.18 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 76
Region of Enrollment [Number; unit: participants]
  Romania | 185

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction of Patients Receiving PegIntron Pen Plus Rebetol Therapy, Assessed by a Survey.
Description: The scale used in the patient questionnaire ranged from 0 (dissatisfied) to 8 (very satisfied). Patients evaluated the training received from the medical staff, ease of the preparation and administration of the medication, and the personal experience when using the PegIntron pen.
Time Frame: The survey was administered during a follow-up visit in the clinic, at any point during the 48-week treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Treated Patients
Number analyzed (Participants) | 182
Units on a scale | 6.16 (0.96)

ADVERSE EVENTS:
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 0/183
Other Adverse Events (participants affected / at risk) | 14/183
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=183)
Pyrexia (General disorders) | 14 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No